CLINICAL TRIAL: NCT06796244
Title: Effectiveness of the Croq'Santé Nutrition Education Program in Improving Food Literacy in Schoolchildren: a Controlled Before-and-after Study in France
Brief Title: Effectiveness of the Croq'Santé Nutrition Education Program in Improving Food Literacy in Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie HERR (Other)
Responsible Party: Sponsor-Investigator, Marie HERR, Professor of Public Health, University of Versailles
Organization: University of Versailles (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UVersailles
Record Dates: First submitted 2025-01-17; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Obesity Prevention; Cancer Prevention
Keywords: food literacy; school-based intervention; nutrition education; prevention program; health promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Schools receiving the Croq'Santé program
  Interventions: Other: Croq'Santé nutrition education program
- Control (No Intervention): Schools delivering usual nutrition education

INTERVENTIONS:
Other: Croq'Santé nutrition education program — The Croq'Santé program aims to develop food literacy in children aged 8 to 11 years. It is based on the creation or adaptation of a recipe chosen by the children. The program is designed to run over the course of one school year, with approximately ten sessions. These sessions are delivered in schools by teachers, following a 3-hour training course. Teachers receive an intervention kit that includes a guide for conducting the different sessions, food images, and a mascot, which children can accessorize as they complete sessions and challenges. The sessions are organized around four stages: discover, invent, cook, and taste. Challenges are to be completed at the end of each stage with the child's family. At the end of the program, children are invited to cook and taste their recipe in a dedicated environment.
  Arms: Intervention

SUMMARY:
Background: Nutritional factors including diet, physical activity, weight status and alcohol consumption are among the most important preventable risk factors for cancer. Interventions are needed to help children make the right choices in a complex food environment. The JDB Foundation designs primary cancer prevention projects through health education targeted at young people. It has designed the "Croq'Santé" project, which aimed to reduce the risks associated with overweight and obesity by improving food literacy of children aged 8 to 11, corresponding to the 4th and 5th grades. Briefly, food literacy refers to having the knowledge, skills and attitudes to choose, prepare and enjoy healthy foods. Accompanied by their teacher, a class will create a balanced recipe (or re-adapt an existing one) through a series of stages (10 sessions in total), allowing children to explore the foods and stakeholders in the food chain, understand nutrition, cook and taste new flavors. Objectives: The primary objective of this study is to evaluate whether the intervention successfuly improves the food literacy of 8- to 11-year-olds. Secondary objectives include examining the influence of socioeconomic factors on the program's effectiveness and process evaluation. Methods: We intent to conduct a quasi-experimental before-and-after study including 60 classes (approximately 1500 children). The classes in the intervention group will receive the Croq'Santé program, while the classes in the control group will receive usual school nutrition education. The schools participating in the control group will have the possibility to receive the Croq'Santé program the following year if they wish. The primary outcome will focus on changes in food literacy, measured using a child-friendly questionnaire administered before and after the intervention. Other information will be collected at child level (e.g. gender, age, family composition) and school level (e.g. socioeconomic indicators). Expected results: Cancer remains the leading cause of death in France and the production of knowledge on the effectiveness of public health interventions is essential to guide prevention strategies. If the Croq'Santé programme actually shows its effectiveness, it could be scaled up and adapted to different contexts.

ELIGIBILITY:
Inclusion Criteria:

* children in 4th and 5th grades
* attending a school participating in the study
* child and parental consent

Exclusion Criteria:

- classes that took part in the questionnaire pre-test

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1205 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Food literacy | The food knowledge questionnaire was administered before the start of the program and at the end of the program, i.e. up to 6 months after the first administration.
  Food literacy was assessed using a score (ranging from 0 to 25, the higher the better) computed from 25 items covering cooking skills, food and nutrition knowledge, attitude towards food, and eating habits (Dallant, Appetite 2024).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation JDB Prévention cancer, Fontenay-lès-Briis, France

IPD SHARING:
Plan to Share IPD: No
The data collected in this study are intended for the evaluation of the Croq'Santé program.